CLINICAL TRIAL: NCT02267954
Title: What's Wrong With This Photo? Fast Food Literacy Study
Brief Title: Fast Food Photo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Eric VanEpps, PhD Candidate, Carnegie Mellon University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS14-582
Record Dates: First submitted 2014-10-14; First posted 2014-10-20 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Calories; Fast Food Literacy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50% Prices/50% Calories (Experimental): The participant is exposed to the baseline menu, but the prices are edited to be at 50% of the actual price (e.g., a $1 coffee is listed as costing $.50) and the calorie labels are edited to be at 50% of the actual content (e.g., a 500 calorie Large Fries is listed as having 250 calories). In addition, the baseline mistakes are still included.
  This is the "Menu edited" intervention.
  Interventions: Other: Menu edited

INTERVENTIONS:
Other: Menu edited — The menu is edited to change price label to 50% of actual value and calorie label to 50% of the actual value, along with other changes.
  Other Names: 50% Prices/50% Calories

SUMMARY:
The investigators aim to discover if people of different demographic levels are more or less attentive to changes in calorie information vs. changes in price information on a restaurant menu. The investigators will record whether the calorie/price change was noticed or not, as well as how quickly the calorie/price change was noticed, depending on condition and individual differences.

DETAILED DESCRIPTION:
Participants complete a short study regarding their ability to detect "mistakes" in a printed version of a fast food restaurant menu. We ask participants to identify the differences between the menu board and a typical menu board at that location. Individuals list the differences that they find and have a chance to win a prize if they identify the most mistakes among participants recruited that day. The differences created will remain constant (e.g., featuring Pepsi products instead of the typical Coca-Cola offerings, including items from other restaurants on the menu), including changes to calorie labels and price labels. Additionally, we recruit participants in a variety of locations to test for differences between demographics (e.g., income groups, education levels, and BMI levels).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Speaks English
* Willing to complete both task and follow-up survey

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Calorie and Price Mistakes Noticed | 10 minutes
  Did participants indicate that a mistake was present in the calorie labels or price labels?

SECONDARY OUTCOMES:
Time until Calorie and Price Mistakes Noticed | 10 minutes
  How long in seconds did it take before participants indicated that a mistake was present in the calorie labels or price labels?
Mistake Number for Calorie and Price Mistakes Noticed | 10 minutes
  How many other mistakes were noticed before calorie/price mistake was noticed?

CONTACTS AND LOCATIONS:
Overall Officials: Eric M VanEpps, MS, Principal Investigator — Carnegie Mellon University
Locations (2):
- United States (2):
  - Community College of Allegheny County, Pittsburgh, Pennsylvania
  - Carnegie Mellon University, Pittsburgh, Pennsylvania